CLINICAL TRIAL: NCT03810443
Title: Prevalence of the Hyperventilation Syndrome in Pulmonary Arterial Hypertension
Acronym: HYPER2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180352
Record Dates: First submitted 2018-12-20; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Hyperventilation
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hyperventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulmonary arterial hypertension (Experimental): The elements of the research consist of the Nijmegen questionnaire response, two dyspnea questionnaires (Dyspnea 12, MDP), a quality of life questionnaire (SF36), a psychological disorder screening questionnaire (HAD) and a diagnostic test: the hyperventilation test.
  Interventions: Diagnostic Test: Hyperventilation test

INTERVENTIONS:
Diagnostic Test: Hyperventilation test — The elements of the research consist of the Nijmegen questionnaire response, two dyspnea questionnaires (Dyspnea 12, MDP), a quality of life questionnaire (SF36), a psychological disorder screening questionnaire (HAD) and a diagnostic test: the hyperventilation test.
  Other Names: Questionnaire of Nijmegen; Questionnaire of Dyspnea; Questionnaire of quality of life; Questionnaire of screening for psychological disorders

SUMMARY:
Dyspnea is a major symptom in pulmonary arterial hypertension and people with the same haemodynamic have generally different degree of dyspnea in pulmonary arterial hypertension. The hyperventilation syndrome is a frequent cause of dyspnea in general population and in respiratory diseases like asthma but has never been studied in pulmonary hypertension. The goal of this study is to measure the prevalence of pulmonary hypertension in a population of patients with controlled pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
Hyperventilation syndrome has been described as a cause of dyspnea in the general population and in several chronic respiratory diseases such as asthma with 20 to 40% of asthmatics affected. However, Hyperventilation syndrome has never been sought in a population with PAH. Hyperventilation syndrome, although complex pathophysiology, may be simply corrected by a management of respiratory physiotherapy based on the control of respiration.

ELIGIBILITY:
Inclusion Criteria:

* Non smoker or tobacco stopped for minimum 2 years ans maximum 10 year-pack. - Idiopathic, heritable, related to drug or toxics, associated with controlled pulmonary hypertension. Diagnosis and treatment of pulmonary hypertension for more than 4 months.
* Optimal control of pulmonary hypertension (no right heart failure symptom and NTproBNP < 300ng/L or Brain Natriuretic Peptide(BNP) < 50 ng/L and optimal hemodynamic results measured by a right heart catheterization in the last year: right atrial pressure < 8 mmHg, cardiac index > 2,5 L/min/m2, veinous saturation in oxygen > 65%)
* Informed and written consent
* Non-affiliation to a social security

Exclusion Criteria:

* Existence of another form of pulmonary hypertension
* Existence of vocal cord dysfunction
* Pregnancy
* Obesity> stage 2 (BMI 35 kg / m2)
* Age ≥ 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-14 (Estimated); Primary Completion 2021-07-14 (Estimated); Study Completion 2021-07-14 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the hyperventilation syndrome | 18 months
  Prevalence of the hyperventilation syndrome in a population with pulmonary arterial hypertension

SECONDARY OUTCOMES:
anxiety-depression questionary score | 18 months
  results of anxiety-depression questionary
dyspnea score | 18 months
  results of dyspnea questionary
quality of life score | 18 months
  results of quality of life questionary

CONTACTS AND LOCATIONS:
Overall Officials: Etienne-Marie JUTANT, CCA, Principal Investigator — APHP
Locations (1):
- Hôpital Bicêtre - Pneumology department, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No